CLINICAL TRIAL: NCT04198376
Title: The Laterally Closed Tunnel Versus Modified Coronally Advanced Tunnel With Subepithelial Connective Tissue Graft for Treatment of Deep Isolated Mandibular Anterior Gingival Recession Defects: A Randomized Controlled Clinical Trial
Brief Title: The Laterally Closed Tunnel Versus Modified Coronally Advanced Tunnel for Mandibular Anterior Gingival Recession Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_91555
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The patients will be assigned into two treatment groups Group A (Test Group) comprises of patient undergoing The Laterally Closed Tunnel Technique with SCTG and Group B(Control Group) comprises of patients undergoing Modified Coronally Advanced Tunnel Technique with SCTG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Laterally Closed Tunnel Technique with SCTG (Experimental): Following the administration of local anaesthesia 2% lignocaine hydrochloride.In the LCT technique a bevelled intrasulcular incisions will be made around the necks of the affected teeth with Orban Knife.The tunnelling will be accomplished with tunneling instrument (TKN2).A mucoperiosteal tunnel will be prepared using a specially designed tunneling instrument.The muscle and collagen fibres will be released using surgical blades and gracey curettes. Subepithelial CTG will be harvested from palate using single incision technique.The graft will be removed and will be placed on saline soaked gauze and kept wet until its transfer to the recipient bed.An immediate closure of the donor site is performed using modified mattress sutures.The graft will be adapted to the CEJ by means of sling suture.Finally the margins of the pouch will be pulled together over the graft and sutured with interrupted sutures
  Interventions: Procedure: Group A The Laterally Closed Tunnel Technique with SCTG
- Modified Coronally Advanced Tunnel Technique with SCTG. (Experimental): In MCAT technique all the buccal tissues will be undermined and connected only the papillary region will be left attached.A full thickness preparation of the papillary region will be created this will be done with a small elevator .A second surgical site will be prepared to obtain the subepithelial CTG using single incision technique.A support suture will be performed to guide the CTG into the recipient site. After sutures are slid through each tunnelled interdental area the needle will be pushed through the CTG before it is guided back through the undermined tissues.The graft will be gently pushed into the pouch with a packing instrument and by pulling the support suture.The entire gingival papillary complex will be moved coronally using a vertical mattress suture anchored in the lingual gingiva.The anchorage in the lingual gingiva will be placed far apically.The suture must capture the buccal flap and graft to avail optimal stabilization.
  Interventions: Procedure: Group B Modified Coronally Advanced Tunnel Technique with SCTG.

INTERVENTIONS:
Procedure: Group A The Laterally Closed Tunnel Technique with SCTG — Following the administration of local anaesthesia 2% lignocaine hydrochloride.In the LCT technique a bevelled intrasulcular incisions will be made around the necks of the affected teeth with Orban Knife.The tunnelling will be accomplished with tunneling instrument (TKN2).A mucoperiosteal tunnel will be prepared using a specially designed tunneling instrument.The muscle and collagen fibres will be released using surgical blades and gracey curettes.Subepithelial CTG will be harvested from palate using single incision technique.The graft will be removed and will be placed on saline soaked gauze and kept wet until its transfer to the recipient bed.An immediate closure of the donor site is performed using modified mattress sutures.The graft will be adapted to the CEJ by means of sling suture.Finally the margins of the pouch will be pulled together over the graft and sutured with interrupted sutures.The surgical sites will be protected with a non eugenol periodontal dressing.
  Arms: The Laterally Closed Tunnel Technique with SCTG
Procedure: Group B Modified Coronally Advanced Tunnel Technique with SCTG. — In MCAT technique all the buccal tissues will be undermined and connected only the papillary region will be left attached.A full thickness preparation of the papillary region will be created this will be done with a small elevator.A second surgical site to obtain the subepithelial CTG using single incision technique.A support suture will be performed to guide the CTG into the recipient site.The graft will be gently pushed into the pouch with a packing instrument and by pulling the support suture.The entire gingivopapillary complex will be moved coronally using a vertical mattress suture anchored in the lingual gingiva.The anchorage in the lingual gingiva will be placed far apically.The suture must capture the buccal flap and graft to avail optimal stabilization.The surgical sites will be protected with a non eugenol periodontal dressing.
  Arms: Modified Coronally Advanced Tunnel Technique with SCTG.

SUMMARY:
The aim of this study is to comparatively evaluate the advantages of LCT with SCTG over MCAT with SCTG for coverage of deep isolated mandibular anterior recession.

DETAILED DESCRIPTION:
Gingival recession is defined as the displacement of the soft tissue margin apical to the cementoenamel junction.Different predisposing anatomic features can result in recession such as position and anatomy of teeth in the dental arch, bony dehiscence, thickness of the alveolar mucosa, muscle pull, orthodontic treatment, thin gingival biotype, buccal prominence of teeth, lack of keratinized tissue, high frenum attachment, or patient related factors such as vigorous brushing or chronic gingival inflammation.

It is a common finding in patient with a high standard of oral hygiene as well as in periodontally untreated populations with poor oral hygiene.The migration of the marginal tissue to an apical position may lead to esthetic concern, dentin hypersensitivity, root caries, and cervical wear.

Mandibular gingival recession defects present significant therapeutic challenges such as shallow vestibular depth, high frenal attachment, thin soft tissue biotypes leading to thin coronally advanced flaps, and thin often dehisced labial bone.Due to these factors the mandibular sites suffers strong and constant tension in comparison to the maxilla, hence there is lack of predictability in the mandibular sites.

Various surgical techniques have been proposed for the treatment of isolated mandibular recessions including the use of fully or partially epithelized free gingival grafts (FGG) or sub epithelial connective tissue graft in conjunction with various types of flaps eg: (envelope, coronally or laterally positioned flap, double pedicle flap (DPF) or tunnelling (TUN) alone or combined with laterally positioned pedicle flaps (LPPF).

Coronally advanced flap (CAF) +connective tissue graft (CTG) is considered as the gold standard treatment in reducing or eliminating gingival recession. Tunnel technique was first introduced by Allen in 19949, and its modifications by Zabalegui in 199910, Modified Coronally Advanced Tunnel (MCAT) by Azzi et al 2002 and Microsurgical CAT by Zuhr 2007.

However, in deep isolated mandibular recessions located in the anterior area, tension free coronal displacement of the flap can be extremely difficult and may result in decreased vestibular depth and flap dehiscence due to increased flap tension.

Therefore a new clinical approach of The Laterally Closed Tunnel (LCT), specifically designed for deep isolated anterior Mandibular Millers class I, II and III recession has been introduced to predictably cover recession and minimize the risk for post operative complications caused by unfavourable anatomical situations.

The important aspect of LCT is the wide mesiodistal and apical mobilisation of the tunnel which enables tension free lateral movement of the flap margins to cover the graft and the recession. The tension free lateral movement and the passive lateral closure of the tunnel margins maybe advantageous in the treatment of isolated deep recessions located in areas with inserting frenula or shallow vestibule, which makes a coronal tension free advancement of the flap extremely difficult.

Beside the tension free flap preparation, the use of SCTG plays a key role in increasing flap thickness and blood clot stability and in providing the cells needed for soft tissue regeneration and keratinization.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Miller's class I, II, III or combined recession defects in mandibular arch.
* Age >/= 18 years.
* Patients with healthy or treated periodontal conditions.
* Patients willing to participate in the study.
* Absence of uncontrolled medical conditions.
* Full mouth plaque score </= 10%(O'Leary 1972).
* Full mouth bleeding score <10%(Ainamo and Bay 1975).
* Patients with esthetic concerns.

Exclusion Criteria:

* Pregnant or lactating females.
* Tobacco smoking.
* Uncontrolled medical conditions.
* Untreated periodontal conditions.
* Use of systemic antibiotics in the past 3 months.
* Patients treated with any medication known to cause gingival hyperplasia.
* Drug and alcohol abuse.
* No occlusal interferences.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Gingival Recession Depth (RD) | 6 Months
  measured as the distance from the CEJ to the gingival margin.

SECONDARY OUTCOMES:
Complete Root Coverage (CRC). | 6 Months
  At 6 months follow up the complete root coverage for control and test group were calculated in % , each group having 12 participants each.
Mean Root Coverage (MRC) | 6 Months
  The mean root coverage % achieved in control group and test group at baseline, 3 months and 6 months with each group having 12 participants each
Gingival Biotype Thickness | 6 Months
  Measured 3mm apically from the free gingival margin at the mid buccal aspect of the tooth.
Apico-coronal Width of Keratinized Tissue (KTW) | 6 Months
  measured as the distance from the mucogingival junction to the gingival margin, with the mucogingival junction location determined using a visual method with Schiller's Potassium Iodide Solution
Root coverage Esthetic Score (RES) | 6 Months
  Cairo 2009
  The RES system evaluated five variables 6 months following surgery: GM, marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment,and gingival color (GC)
  GM.Zero points=failure of root coverage (gingival margin apical or equal to the baseline recession); 3points=partial root coverage; 6 points=CRC MTC.Zero points=irregular gingival margin (doesnot follow the CEJ); 1 point=proper marginal contour/scalloped gingival margin (follows the CEJ).
  STT.Zero points=scar formation and/or keloid-like appearance; 1 point=absence of scar or keloid formation MGJ.Zero points=MGJ not aligned with the MGJ of adjacent teeth; 1 point=MGJ aligned with the MGJ of adjacent teeth.
  GC.Zero points=color of tissue varies from gingival color at adjacent teeth; 1 point=normal color and integration with the adjacent soft tissues.
  The ideal esthetic score was 10.
Gingival Recession Width | 6 Months
  Measured as the distance between the mesial gingival margin and distal gingival margin
Pocket Probing Depth | 6 Months
  Measured as the distance from the gingival margin to the base of gingival sulcus
Clinical Attachment Level | 6 Months
  Measured as Gingival Recession Depth+Probing Depth
Plaque Index (PI) | 6 Months
  Silness and Loe 1964
  PI=0 score given when the gingival area of the tooth surface is literally free of plaque.
  PI=1 represents the situation where the gingival area is covered with a thin film of plaque which is not visible,but which is made visible PI=2 score given when the deposit is visible PI=3 is reserved for the heavy (1-2mm.thick) accumulation of soft matter.
Gingival Index (GI) | 6 Months
  Loe and Silness 1963
  The criteria are: 0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
  A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation
Bleeding Index (BI) | 6 Months
  Ainamo and Bay 1975 It is performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Phebie Asta Rodrigues, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences; Dr.Joann Pauline George, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karantaka, India

IPD SHARING:
Plan to Share IPD: No